CLINICAL TRIAL: NCT02304003
Title: The Effect of an Evidence-based Physiotherapy Regimen for Patients on Need for Subacromial Decompression Surgery Due to Rotator Cuff Tendinopathy : a Randomized Controlled Trial.
Brief Title: The Effect of an Evidence-based Physiotherapy Regimen for Patients With Rotator Cuff Tendinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bergen University College (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Principal Investigator, Sturla Haslerud, Sturla Haslerud , PT , Msc Orthopedics & Reumatology , PhD candidate, Bergen University College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BergenUC; 2012/2134 (Other: Regional Ethics Committee Norway , REK Nord)
Record Dates: First submitted 2014-11-26; First posted 2014-12-01 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Tendinopathy; Shoulder Impingement Syndrome; Shoulder Pain; Subacromial Impingement
Keywords: Shoulder tendinopathy; Subacromial impingement syndrome; Rotator cuff tendinopathy; Supraspinatus tendinopathy
MeSH Terms: conditions — Tendinopathy; Shoulder Impingement Syndrome; Shoulder Pain | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Structured Physiotherapy regimen (Experimental): Heavy-slow resistance training of rotator cuff . Scapular exercises. Manual mobilisation of glenohumeral joint . Stretching. Low Level Laser therapy
  Interventions: Other: Structured Physiotherapy Regimen
- Standard care (Other): Standard care offered in primary care while waiting for surgery , this may be but are not limited to : Wait and see, Drugs ( NSAIDS ), Corticosteroid injections, physiotherapy or other conservative treatment options.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Structured Physiotherapy Regimen — Experimental group will be treated with heavy-slow resistance exercises targeted at the rotator cuff tendons, and exercises to improve scapular stability and strength. Glenohumeral mobilisation techniques and and stretching of glenohumeral capsule and pectoralis minor. Rotator cuff tendons and glenohumeral synovia will be irradiated with low level laser according to WALT dosage recommendations . Intervention period is 12 weeks. Three weekly treatment sessions at 0-3 weeks. 4-12 weeks one treatment session weekly , and two days of home-exercise per week.
  Arms: Structured Physiotherapy regimen
Other: Standard Care — Standard follow up in primary care.
  Arms: Standard care

SUMMARY:
Primary aim of this study is to investigate wether an evidence-based physiotherapy regimen is more effective than standard care in patients referred for arthroscopic surgery of the shoulder. It is hypothesized that a multimodal physiotherapy regimen will relieve pain, improve shoulder function and reduce the need for subacromial decompression surgery of the shoulder compared to standard care/wait and see controls.

DETAILED DESCRIPTION:
There has been a fourfold increase in surgery rates for non-traumatic shoulder disorders , despite increasing evidence demonstrating that there is no difference in effect between physiotherapy based- and surgical interventions. The target population for this study is patients suffering from rotator cuff tendinopathy waiting for subacromial decompression surgery at a university hospital in Norway. During this waiting period , study participants will be randomly assigned to standard follow up or a physiotherapy regimen in primary care. We want to compare the effect of a structured physiotherapy regimen consisting of heavy slow resistance exercises, stretching, manual mobilization and low level laser therapy to standard follow up.

ELIGIBILITY:
Inclusion Criteria:

Patients on need for surgery ( placed at surgical waiting list at hospital or referred to surgery by their GP )

1. Typical history with difficulties working with arms elevated over the head, and pain located in the upper segment of C5 dermatome.
2. Symptom duration of minimum 3 months.
3. Three or more reproducible signs of rotator cuff tendinopathy / subacromial impingement:

   * Positive isometric abduction and/or lateral rotation (Ombregt, Bisschop & Veer, 2003)
   * Painful arc during active abduction (Ombregt, Bisschop & Veer, 2003)
   * Positive Neers sign (Neer, 1972 ; Tennent, Beach & Meyers, 2003)
   * Positive Jobes test (Jobe & Moynes, 1982 ; Tennent, Beach & Meyers, 2003)
   * Positive Hawkins-Kennedy impingement test (Hawkins & Kennedy, 1980)

Exclusion Criteria:

1. Shoulder pain due to trauma, e.g. fall.
2. Reduced ROM consistent with adhesive capsulitis/frozen shoulder
3. History in combination with examination and tests (apprehension/relocation), giving reason to suspect pathological instability
4. Full thickness rupture of rotator cuff tendon
5. OA of the glenohumeral joint, Os acromiale with decreased space of the subacromial space, previous fractures in the shoulder complex or shoulder surgery on the symptomatic side.
6. Subjects with other comorbidity: Rheumatological or neurological disease, fibromyalgia or symptoms from the cervical spine
7. Subjects suffering from serious psychiatric illness.
8. Subjects unable to understand English or Norwegian.
9. Less than 3 positive reproducible sings of rotator cuff pathology / subacromial disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Need for surgery | 12 weeks (end of treatment) and 6 months post treatment
  Dichotomised questionnaire yes or no
Shoulder function | 4 weeks , 12 weeks and 6 months
  Shoulder Pain and Disability Index. 13 questions. To answer the questions, patients place a mark on a 10 point numerical scale for each question. Verbal anchors for the pain dimension are 'no pain at all' and 'worst pain imaginable', and those for the functional activities are 'no difficulty' and 'so difficult it required help'.
Shoulder Pain | 4 weeks , 12 weeks and 6 months
  Night pain assessed on a 10 point numerical scale . Pain now and this week measured on a 10 point numerical scale .
Generic health status | 12 weeks and 6 months
  EQ-5D questionaire. The system comprises the following 5 dimensions: mobility, self-care, usual activities,pain and anxiety/depression. he respondent is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions.

SECONDARY OUTCOMES:
Rotator cuff force | 12 weeks ( end of treatment)
  Maximal painfree isometric force measurements of rotator cuff muscles using handheld dynamometry .
Tendon pain pressure threshold | 12 weeks ( end of treatment )
  Tendon pressure applied over individual rotator cuff tendons with analogue algometer. Pain threshold registered in kilograms.
Analgesics and corticosteroid injections | 4 weeks , 12 weeks and 6 months
  Analgesics consumption and corticosteroids injections registered on questionaire.
Tendon thickness | 12 weeks ( end of treatment )
  Ultrasonography measurements of rotator cuff tendon thickness ( subscapularis , supraspinatus , infraspinatus , biceps )
Patient global impression of change | 4 weeks, 12 weeks & 6 months
  To assess global improvement a 7 point categorical scale ranging from " much better to much worse" is used.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Magnus Bjordal, Professor, Study Chair — University of Bergen , Dep. of Global Public Health and Primary Care, Physiotherapy Research Group, Norway.
Locations (1):
- Department of Physiotherapy, Hillevaag General Practitioner Practice, Stavanger, Norway